CLINICAL TRIAL: NCT01532869
Title: A Phase II/III, Multicenter, Randomized, Double-blind, Placebo-controlled Study To Assess The Efficacy And Safety Of Tocilizumab Versus Placebo In Patients With Systemic Sclerosis
Brief Title: A Study of RoActemra/Actemra (Tocilizumab) Versus Placebo in Patients With Systemic Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WA27788; 2011-001460-22 (EudraCT Number)
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Results first posted 2015-11-05 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-08

CONDITIONS: Sclerosis, Systemic
MeSH Terms: conditions — Scleroderma, Systemic | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: tocilizumab [RoActemra/Actemra]
- Tocilizumab (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: Placebo — Subcutaneously weekly, Weeks 0-48
  Arms: Placebo
Drug: tocilizumab [RoActemra/Actemra] — 162 mg subcutaneously weekly, Weeks 0-48
  Arms: Tocilizumab
Drug: tocilizumab [RoActemra/Actemra] — 162 mg subcutaneously weekly, Week 48-96

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled, two-arm, parallel-group study will evaluate the efficacy and safety of RoActemra/Actemra (tocilizumab) in participants with systemic sclerosis. Participants will be randomized to receive either RoActemra/Actemra 162 mg subcutaneously weekly or placebo for 48 weeks. From Week 48 to Week 96, all participants will receive open-label RoActemra/Actemra 162 mg subcutaneously weekly. Anticipated time on study treatment is 96 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Systemic sclerosis, as defined by American College of Rheumatology (1980) criteria
* Disease duration of </= 60 months (defined as time from first non-Raynaud phenomenon manifestation)
* >/= 15 and </= 40 mRSS units at screening
* Active disease, as defined by protocol
* Uninvolved skin at injection sites
* Negative pregnancy test for a female subject of childbearing potential

Exclusion Criteria:

* Major surgery (including joint surgery) within 8 weeks prior to and/or during study enrollment
* Rheumatic autoimmune disease other than systemic sclerosis
* Skin thickening (scleroderma) limited to areas distal to the elbows or knees at screening
* Previous treatment with tocilizumab
* History of severe allergic or anaphylactic reactions to human, humanized, or murine monoclonal antibodies
* Severe cardiopulmonary disease
* Known active current or history of recurrent infections
* Use of any investigational, biologic, or immunosuppressive therapies including intra-articular or parenteral corticosteroids prior to study enrollment as specified in the protocol
* As specified in the protocol, any current or past medical condition or medical history involving but not limited to the nervous, renal, pulmonary, endocrine, and gastrointestinal organ systems determined by the Principal Investigator to pose a significant safety risk to any subject while participating in the study
* Primary or secondary immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (50):
- United States (21):
  - Los Angeles, California
  - San Diego, California
  - Stanford, California
  - Farmington, Connecticut
  - Washington D.C., District of Columbia
  - Chicago, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - New Brunswick, New Jersey
  - Lake Success, New York
  - New York, New York
  - Cleveland, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Charleston, South Carolina
  - Houston, Texas
  - Salt Lake City, Utah
  - Seattle, Washington
- Canada (3):
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
- France (6):
  - Bordeaux
  - Caen
  - Lille
  - Paris
  - Strasbourg
  - Toulouse
- Germany (11):
  - Bad Nauheim
  - Baden-Baden
  - Berlin
  - Bochum
  - Cologne
  - Dresden
  - Erlangen
  - Frankfurt
  - Hamburg
  - Tübingen
  - Ulm
- United Kingdom (9):
  - Cannock
  - Dundee
  - Edinburgh
  - Leeds
  - Liverpool
  - London
  - Middlesbrough
  - Newcastle upon Tyne
  - Romford

REFERENCES:
- [Derived] Gao X, Jia G, Guttman A, DePianto DJ, Morshead KB, Sun KH, Ramamoorthi N, Vander Heiden JA, Modrusan Z, Wolters PJ, Jahreis A, Arron JR, Khanna D, Ramalingam TR. Osteopontin Links Myeloid Activation and Disease Progression in Systemic Sclerosis. Cell Rep Med. 2020 Nov 17;1(8):100140. doi: 10.1016/j.xcrm.2020.100140. eCollection 2020 Nov 17. PMID 33294861
- [Derived] Stifano G, Sornasse T, Rice LM, Na L, Chen-Harris H, Khanna D, Jahreis A, Zhang Y, Siegel J, Lafyatis R. Skin Gene Expression Is Prognostic for the Trajectory of Skin Disease in Patients With Diffuse Cutaneous Systemic Sclerosis. Arthritis Rheumatol. 2018 Jun;70(6):912-919. doi: 10.1002/art.40455. PMID 29858547
- [Derived] Denton CP, Ong VH, Xu S, Chen-Harris H, Modrusan Z, Lafyatis R, Khanna D, Jahreis A, Siegel J, Sornasse T. Therapeutic interleukin-6 blockade reverses transforming growth factor-beta pathway activation in dermal fibroblasts: insights from the faSScinate clinical trial in systemic sclerosis. Ann Rheum Dis. 2018 Sep;77(9):1362-1371. doi: 10.1136/annrheumdis-2018-213031. Epub 2018 May 31. PMID 29853453
- [Derived] Khanna D, Denton CP, Lin CJF, van Laar JM, Frech TM, Anderson ME, Baron M, Chung L, Fierlbeck G, Lakshminarayanan S, Allanore Y, Pope JE, Riemekasten G, Steen V, Muller-Ladner U, Spotswood H, Burke L, Siegel J, Jahreis A, Furst DE. Safety and efficacy of subcutaneous tocilizumab in systemic sclerosis: results from the open-label period of a phase II randomised controlled trial (faSScinate). Ann Rheum Dis. 2018 Feb;77(2):212-220. doi: 10.1136/annrheumdis-2017-211682. Epub 2017 Oct 24. PMID 29066464
- [Derived] Khanna D, Denton CP, Jahreis A, van Laar JM, Frech TM, Anderson ME, Baron M, Chung L, Fierlbeck G, Lakshminarayanan S, Allanore Y, Pope JE, Riemekasten G, Steen V, Muller-Ladner U, Lafyatis R, Stifano G, Spotswood H, Chen-Harris H, Dziadek S, Morimoto A, Sornasse T, Siegel J, Furst DE. Safety and efficacy of subcutaneous tocilizumab in adults with systemic sclerosis (faSScinate): a phase 2, randomised, controlled trial. Lancet. 2016 Jun 25;387(10038):2630-2640. doi: 10.1016/S0140-6736(16)00232-4. Epub 2016 May 5. PMID 27156934

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization was stratified by joint involvement at baseline (>=4 or <4 tender joints of 28 tender joint count [TJC]). The study consisted of double-blind (Week 0-Week 48) and open-label (Week 48-Week 96) periods. Data analyzed up to Weeks 24 and 48 (data cut-off: 11 July 2014), and up to Week 96 (data cut-off: 05 August 2015) are reported.
Groups:
- Placebo: Participants received tocilizumab (TCZ) matched placebo by subcutaneous (SC) injection every week (qw) for Week 0 to Week 48 (blinded-treatment period) and then received TCZ (162 milligrams [mg]) SC injection qw in the open-label period for Week 48 to Week 96.
- Tocilizumab: Participants received TCZ (162 mg) by SC injection qw for Week 0 to Week 48 (blinded-treatment period) and then in the open-label period for Week 48 to Week 96.
Period: Blinded-Treatment Period (Up to Week 24)
Arm/Group | Placebo | Tocilizumab
Started | 44 | 43
Completed | 36 (Number of participants who completed the first 24 weeks of full 48 weeks blinded-treatment period.) | 35 (Number of participants who completed the first 24 weeks of full 48 weeks blinded-treatment period.)
Not Completed | 8 | 8
Not completed — Death | 0 | 1
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliance | 1 | 0
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 4 | 2
Period: Blinded-Treatment Period (Up to Week 48)
Arm/Group | Placebo | Tocilizumab
Started | 44 | 43
Completed | 33 (Number of participants who completed 48 weeks of blinded-treatment period.) | 30 (Number of participants who completed 48 weeks of blinded-treatment period.)
Not Completed | 11 | 13
Not completed — Death | 0 | 3
Not completed — Adverse Event | 4 | 5
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-Compliance | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Physician Decision | 1 | 0
Period: Open-label Period (Week 48 to Week 96)
Arm/Group | Placebo | Tocilizumab
Started | 31 (Two participants did not start the open label extension period.) | 30
Completed | 24 (Number of participants who completed study to Week 96.) | 27 (Number of participants who completed study to Week 96.)
Not Completed | 7 | 3
Not completed — Adverse Event | 4 | 1
Not completed — Non-compliance | 1 | 0
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received any study drug and provided at least one post-dose safety assessment (withdrawal, adverse event [AE], death, laboratory assessment, vital signs).
Groups:
- Placebo: Participants received TCZ matched placebo by SC injection qw for Week 0 to Week 48 (blinded-treatment period) and then received TCZ (162 mg) SC injection qw in the open-label period for Week 48 to Week 96.
- Total: Total of all reporting groups
Arm/Group | Placebo | Tocilizumab | Total
Number analyzed (Participants) | 44 | 43 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.1 (12.9) | 51.2 (11.7) | 49.6 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Rodnan Skin Score (mRSS) at Week 24
Description: Skin thickness was assessed by the mRSS. The mRSS was rated with scores ranging from 0 (normal) to 3 (severe skin thickening) across 17 different sites. The total score was the sum of the individual skin scores in the 17 body areas (e.g., face, hands, fingers; proximal area of the arms, distal area of the arms, thorax, abdomen; proximal area of the legs, and distal area of the legs, feet), giving a range of 0-51 units and had been validated for participants with systemic sclerosis (SSc). A negative change from baseline showed improvement.
Time Frame: Baseline, Week 24
Population: Intent-to-treat (ITT) population included all participants randomized who had received any study drug at the time of the Week 24 cutoff date (14 January 2014). Here, number of participants analyzed included only those participants who were evaluable for this outcome measure at any time point up to Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: unit on a scale
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 43 | 41
unit on a scale | -1.22 [-3.42 to 0.98] | -3.92 [-6.17 to -1.67]
Statistical Analysis 1: Comparison: Placebo vs Tocilizumab; The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.0915, Mixed Models Analysis; Difference in Least Square (LS) mean = -2.70, 95% CI 2-sided [-5.85 to 0.45]

2. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to Week 8 after last dose that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Week 48
Population: Safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 44 | 43
percentage of participants
  Treatment-emergent adverse events | 90.9 | 97.7
  Treatment-emergent serious adverse events | 34.1 | 32.6

3. Secondary Outcome: Change From Baseline in Physical Function Assessed by Scleroderma Health Assessment Questionnaire Disability Index (SHAQ-DI)
Description: SHAQ-DI assessed five scleroderma-specific visual analogue scale (VAS) items to explore the impact of participant's disease. These items were developed to measure the effect of scleroderma on five elements of disease that could have a great impact on a participant's daily activities. Each VAS item was rated separately (0-100 millimeters [mm]), with higher scores indicating more severe disease. The five items were: 1) intestinal disease, 2) breathing problem, 3) Raynaud syndrome, 4) finger ulcers, and 5) overall disease.
Time Frame: Baseline, Weeks 24 and 48
Population: ITT population. Here, number of participants analyzed included only those participants who were evaluable for this outcome measure and "n" included those who were evaluable for the specific item at specified time point in specified timeframe.
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 42 | 41
mm
  Week 24: Intestinal VAS Score (n=42, 41) | 5.81 [-1.43 to 13.06] | 5.38 [-1.98 to 12.74]
  Week 24: Breathing VAS Scores (n=42, 41) | 8.54 [0.81 to 16.27] | 4.42 [-3.47 to 12.31]
  Week 24: Raynaud syndrome (n=42, 41) | 2.41 [-6.96 to 11.78] | 1.13 [-8.47 to 10.73]
  Week 24: Finger ulcers VAS Score (n=42, 41) | 9.20 [-0.22 to 18.61] | 14.09 [4.45 to 23.73]
  Week 24: Overall disease (n=42, 41) | 1.89 [-4.99 to 8.77] | 1.81 [-5.21 to 8.84]
  Week 48: Intestinal VAS Score (n=41, 41) | 7.91 [-0.37 to 16.18] | 1.11 [-6.88 to 9.10]
  Week 48: Breathing VAS Scores (n=41, 41) | 0.55 [-7.09 to 8.19] | 2.09 [-5.39 to 9.57]
  Week 48: Raynaud syndrome (n=41, 41) | 0.30 [-9.51 to 10.12] | -4.18 [-13.87 to 5.51]
  Week 48: Finger ulcers VAS Score (n=41, 41) | 4.97 [-3.15 to 13.10] | -0.83 [-8.83 to 7.17]
  Week 48: Overall disease (n=41, 41) | 3.46 [-4.50 to 11.41] | -4.36 [-12.27 to 3.55]
Statistical Analysis 1: Comparison: Placebo vs Tocilizumab; Change From Baseline in Intestinal VAS Score at Week 24. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.9336, Mixed Models Analysis; Difference in LS mean = -0.43, 95% CI 2-sided [-10.78 to 9.91]
Statistical Analysis 2: Comparison: Placebo vs Tocilizumab; Change From Baseline in Breathing VAS Score at Week 24. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.4609, Mixed Models Analysis; Difference in LS mean = -4.12, 95% CI 2-sided [-15.21 to 6.96]
Statistical Analysis 3: Comparison: Placebo vs Tocilizumab; Change From Baseline in Raynaud Syndrome Score at Week 24. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.8493, Mixed Models Analysis; Difference in LS mean = -1.28, 95% CI 2-sided [-14.70 to 12.13]
Statistical Analysis 4: Comparison: Placebo vs Tocilizumab; Change From Baseline in Finger Ulcers Score at Week 24. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.4717, Mixed Models Analysis; Difference in LS mean = 4.89, 95% CI 2-sided [-8.59 to 18.37]
Statistical Analysis 5: Comparison: Placebo vs Tocilizumab; Change From Baseline in Overall Disease Score at Week 24. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.9876, Mixed Models Analysis; Difference in LS mean = -0.08, 95% CI 2-sided [-9.93 to 9.78]
Statistical Analysis 6: Comparison: Placebo vs Tocilizumab; Change From Baseline in Intestinal VAS Score at Week 48. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.2407, Mixed Models Analysis; Difference in LS mean = -6.80, 95% CI 2-sided [-18.30 to 4.71]
Statistical Analysis 7: Comparison: Placebo vs Tocilizumab; Change From Baseline in Breathing VAS Score at Week 48. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.7742, Mixed Models Analysis; Difference in LS mean = 1.54, 95% CI 2-sided [-9.18 to 12.26]
Statistical Analysis 8: Comparison: Placebo vs Tocilizumab; Change From Baseline in Raynaud Syndrome Score at Week 48. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.5182, Mixed Models Analysis; Difference in LS mean = -4.48, 95% CI 2-sided [-18.28 to 9.31]
Statistical Analysis 9: Comparison: Placebo vs Tocilizumab; Change From Baseline in Finger Ulcers Score at Week 48. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.3106, Mixed Models Analysis; Difference in LS mean = -5.80, 95% CI 2-sided [-17.20 to 5.59]
Statistical Analysis 10: Comparison: Placebo vs Tocilizumab; Change From Baseline in Overall Disease Score at Week 48. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.1717, Mixed Models Analysis; Difference in LS mean = -7.82, 95% CI 2-sided [-19.11 to 3.48]

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 24 and Week 48
Description: The HAQ-DI scale consisted of 20 questions referring to eight component sets: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. The total score indicated the participant's self-assessed level of disability. There are four possible responses for each component: 0 = without any difficulty; 1 = with some difficulty; 2 = with much difficulty; 3 = unable to do. The HAQ-DI was the sum of the domain scores, divided by the number of domains that have a score (i.e. the average score), with total range of 0 to 3, higher scores showing larger functional limitation.
Time Frame: Baseline, Weeks 24 and 48
Population: ITT population. Here, number of participants analyzed included only those participants who were evaluable for this outcome measure and "n" included those who were evaluable for the specific item at specified time point in specified time frame.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 42 | 41
units on a scale
  Week 24 (n=42, 41) | 0.118 [-0.026 to 0.262] | 0.137 [-0.010 to 0.285]
  Week 48 (n=41, 41) | 0.205 [0.017 to 0.393] | -0.002 [-0.188 to 0.183]
Statistical Analysis 1: Comparison: Placebo vs Tocilizumab; Change From Baseline in HAQ-DI Score at Week 24. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.8503, Mixed Models Analysis; Difference in LS mean = 0.020, 95% CI 2-sided [-0.186 to 0.225]
Statistical Analysis 2: Comparison: Placebo vs Tocilizumab; Change From Baseline in HAQ-DI Score at Week 48. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.1212, Mixed Models Analysis; Difference in LS mean = -0.207, 95% CI 2-sided [-0.471 to 0.056]

5. Secondary Outcome: Change From Baseline in Clinician's Global Assessment at Week 24 and Week 48
Description: The Clinician's Global Assessment evaluated the overall impact of SSc on the participant as assessed by the physician on a VAS with scores ranging from 0 to 100 mm, with higher scores indicating worse disease in terms of severity, damage, or overall disease, but there was no standardization for the scale.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 41 | 40
mm
  Week 24 (n=41, 39) | -7.25 [-12.99 to -1.51] | -8.24 [-14.06 to -2.41]
  Week 48 (n=41, 40) | -9.39 [-16.66 to -2.12] | -18.41 [-25.30 to -11.52]
Statistical Analysis 1: Comparison: Placebo vs Tocilizumab; Change From Baseline in Clinician's Global Assessment at Week 24.The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.8118, Mixed Models Analysis; Difference in LS mean = -0.99, 95% CI 2-sided [-9.20 to 7.23]
Statistical Analysis 2: Comparison: Placebo vs Tocilizumab; Change From Baseline in Clinician's Global Assessment at Week 48.The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.0768, Mixed Models Analysis; Difference in LS mean = -9.02, 95% CI 2-sided [-19.04 to 1.00]

6. Secondary Outcome: Change From Baseline in Patient's Global Assessment at Week 24 and Week 48
Description: The Patient's Global Assessment was a patient's reported outcome that represented the participant's overall assessment of his or her current SSc on a 100 mm horizontal VAS scale (0 mm to 100 mm), with higher scores indicating worsening disease.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 42 | 42
mm
  Week 24 (n=42, 42) | 1.53 [-4.93 to 7.98] | -2.33 [-8.87 to 4.22]
  Week 48 (n=41, 42) | -2.70 [-10.56 to 5.16] | -11.00 [-18.69 to -3.31]
Statistical Analysis 1: Comparison: Placebo vs Tocilizumab; Change From Baseline in Patient's Global Assessment at Week 24. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.4063, Mixed Models Analysis; Difference in LS mean = -3.85, 95% CI 2-sided [-13.04 to 5.34]
Statistical Analysis 2: Comparison: Placebo vs Tocilizumab; Change From Baseline in Patient's Global Assessment at Week 48. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.1371, Mixed Models Analysis; Difference in LS mean = -8.30, 95% CI 2-sided [-19.31 to 2.71]

7. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Score at Week 24 and Week 48
Description: This FACIT-Fatigue Scale was a 13-item measure with participants scoring each item on a 5-point scale (0 to 4) up to 52 points. The endpoint measured was fatigue. On this scale, a numerical increase indicated an improvement in the participant's condition.
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 41 | 42
units on a scale
  Week 24 (n=41, 42) | 1.26 [-1.85 to 4.37] | 2.68 [-0.41 to 5.77]
  Week 48 (n=40, 42) | 0.36 [-2.64 to 3.37] | 3.11 [0.28 to 5.95]
Statistical Analysis 1: Comparison: Placebo vs Tocilizumab; Change From Baseline in FACIT-Fatigue Score at Week 24. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.5197, Mixed Models Analysis; Difference in LS mean = 1.43, 95% CI 2-sided [-2.97 to 5.82]
Statistical Analysis 2: Comparison: Placebo vs Tocilizumab; Change From Baseline in FACIT-Fatigue Score at Week 48. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.1886, Mixed Models Analysis; Difference in LS mean = 2.75, 95% CI 2-sided [-1.38 to 6.88]

8. Secondary Outcome: Change From Baseline in 5-D Itch Scale at Week 24 and Week 48
Description: The 5-D Itch Scale contained five domains of duration, degree, direction, disability, and distribution. The endpoint of the scale was pruritus. Each domain was scored on a 5-point scale, the scores of each of the five domains were achieved separately and then summed together to obtain a total 5-D score. 5-D scores ranged between 5 (no pruritus) and 25 (most severe pruritus).
Time Frame: Baseline, Weeks 24 and 48
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 41 | 41
units on a scale
  Week 24 (n=41, 41) | -1.73 [-2.95 to -0.50] | -0.94 [-2.15 to 0.28]
  Week 48 (n=40, 41) | -1.08 [-2.60 to 0.43] | -2.19 [-3.58 to -0.80]
Statistical Analysis 1: Comparison: Placebo vs Tocilizumab; Change From Baseline in 5-D Itch Scale at Week 24. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.3651, Mixed Models Analysis; Difference in LS mean = 0.79, 95% CI 2-sided [-0.94 to 2.51]
Statistical Analysis 2: Comparison: Placebo vs Tocilizumab; Change From Baseline in 5-D Itch Scale at Week 48. The analysis included the fixed, categorical effects of treatment, visit, the stratification factor of joint involvement at the baseline visit, and treatment-by-visit interaction, as well as the continuous covariates of baseline score and baseline score-by-visit interaction; Test type: Superiority or Other; p = 0.2841, Mixed Models Analysis; Difference in LS mean = -1.11, 95% CI 2-sided [-3.16 to 0.94]

9. Secondary Outcome: Change From Baseline in mRSS at Week 48
Description: as for outcome 1
Time Frame: Baseline, Week 48
Population: ITT population. Here, number of participants analyzed included only those participants who were evaluable for this outcome measure at specified time point up to 48 weeks.
Measure: Least Squares Mean (95% Confidence Interval); unit: unit on a scale
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 43 | 41
unit on a scale | -2.77 [-5.44 to -0.11] | -6.33 [-8.86 to -3.79]
Statistical Analysis 1: Comparison: Placebo vs Tocilizumab; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0579, Mixed Models Analysis; Difference in LS mean = -3.55, 95% CI 2-sided [-7.23 to 0.12]

10. Secondary Outcome: Percentage of Participants Who Maintained or Improved in mRSS From Week 24 to Week 48
Description: Skin thickness was assessed by the mRSS. The mRSS was rated with scores ranging from 0 (normal) to 3 (severe skin thickening) across 17 different sites. The total score was the sum of the individual skin scores in the 17 body areas (e.g., face, hands, fingers; proximal area of the arms, distal area of the arms, thorax, abdomen; proximal area of the legs, and distal area of the legs, feet), giving a range of 0-51 units and had been validated for participants with systemic sclerosis (SSc). A negative change from baseline showed improvement. Percentage of participants with an improvement in mRSS at Week 24 (change from baseline <0) that maintained or further improved at Week 48 were reported as "Yes" and "No" with Yes = improvers at week 24 that had a change from baseline in mRSS at Week 48 <= change from baseline at Week 24.
Time Frame: Week 48
Population: ITT population. Here number of participants analyzed included those with mRSS change from baseline <0 at Week 24 and with non-missing change from baseline in mRSS at Week 48.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 43 | 41
percentage of participants | 44.4 | 68.2
Statistical Analysis 1: Comparison: Placebo vs Tocilizumab; The logistic regression model included the fixed categorical effects of treatment and the stratification factor of joint involvement at the baseline visit. The continuous covariate of baseline mRSS score was also included in the model; Test type: Superiority or Other; p = 0.2159, Regression, Logistic; Odds Ratio (OR) = 2.39, 95% CI 2-sided [0.60 to 9.50], Standard Error of Mean 0.704

11. Secondary Outcome: Change From Baseline in Tender Joint Count 28 (TJC28)
Description: Joint tenderness was evaluated as per assessment of 28 joints. Joints on both sides of the body, including shoulders, elbows, wrists, 10 metacarpal phalangeal (MCP) joints, 10 proximal interphalangeal joint (PIP) joints, and both knees, were assessed. Joints were classified as not tender = 0 or tender = 1. Observed data was presented for this outcome measure.
Time Frame: Baseline, Weeks 3, 8, 16, 24, 32, 40, and 48
Population: ITT population. Here, "n" = participants evaluable for the specific item at specified time point in specified time frame.
Measure: Mean (Standard Deviation); unit: joint count
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 20 | 19
joint count
  Week 3 (n=20, 19) | -2.75 (4.27) | -2.32 (5.55)
  Week 8 (n=18, 19) | -3.06 (6.67) | -4.00 (6.16)
  Week 16 (n=18, 17) | -3.50 (6.00) | -3.65 (7.59)
  Week 24 (n=17, 16) | -2.06 (6.28) | -4.31 (7.34)
  Week 32 (n=12, 11) | -3.33 (6.62) | -3.18 (7.40)
  Week 40 (n=10, 10) | -3.80 (6.76) | -4.30 (8.23)
  Week 48 (n=12, 10) | -2.92 (7.08) | -5.10 (7.29)

12. Secondary Outcome: Area Under the Concentration-Time Curve (AUC) From Time 0 to 168 Hour (AUC0-168)
Description: AUC was a measure of the serum concentration of the drug over time which was measured in micrograms times (*) hour per milliliters (µg*hr/mL). It is used to characterize drug absorption.
Time Frame: Pre-dose, 24, 48, 72, 96, 120 or 144, and 168 hours post dose for Baseline and Week 16
Population: Pharmacokinetic (PK) population included all participants who received at least one TCZ injection and had at least one PK sample with detectable results. Here, "n" = participants evaluable for the specific item at specified time point in specified time frame.
Measure: Mean (Standard Deviation); unit: µg*hr/mL
Arm/Group | Tocilizumab
Number analyzed (Participants) | 7
µg*hr/mL
  Baseline (n=7) | 686 (455)
  Week 16 (n=4) | 7508 (2369)

13. Secondary Outcome: Mean Serum Concentrations of Interleukin (IL)-6 by Visit
Description: Observed data was presented for this outcome measure.
Time Frame: Baseline, Weeks 1, 2, 3, 8, 16, 24, and 48
Population: Safety population. Here, number of participants analyzed included only those participants who were evaluable for this outcome measure and "n" included those who were evaluable for the specific item at specified time point in specified time frame.
Measure: Mean (Standard Deviation); unit: picograms per milliliters (pg/mL)
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 43 | 43
picograms per milliliters (pg/mL)
  Baseline (n=43, 42) | 15.02 (18.19) | 13.57 (14.69)
  Week 1: Absolute values (n=43, 43) | 17.24 (22.77) | 158.91 (326.42)
  Week 1: Change From Baseline (n=42, 42) | 1.33 (27.29) | 147.37 (326.20)
  Week 2: Absolute values (n=43, 41) | 12.60 (13.78) | 107.10 (73.75)
  Week 2: Change From Baseline (n=42, 40) | -3.07 (17.85) | 94.54 (67.99)
  Week 3: Absolute values (n=42, 40) | 12.47 (10.72) | 116.58 (75.31)
  Week 3: Change From Baseline (n=41, 39) | -3.60 (15.28) | 104.44 (71.84)
  Week 8: Absolute values (n=42, 39) | 15.39 (19.04) | 115.31 (66.39)
  Week 8: Change From Baseline(n=41,38) | 0.15 (18.65) | 104.14 (62.95)
  Week 16: Absolute values (n=32,33) | 12.51 (14.06) | 98.36 (61.65)
  Week 16: Change From Baseline (n=31,32) | -1.26 (11.34) | 88.86 (59.77)
  Week 24: Absolute values (n=36,34) | 10.19 (10.55) | 84.67 (68.37)
  Week 24: Change From Baseline(n=35,33) | -2.74 (12.43) | 73.61 (68.07)
  Week 48: Absolute values (n=32,27) | 10.50 (11.82) | 65.30 (35.95)
  Week 48: Change From Baseline (n=31,26) | -2.61 (14.92) | 55.60 (35.86)

14. Secondary Outcome: Mean Serum Concentrations of Soluble IL-6 Receptor (R) by Visit
Description: Observed data was presented for this outcome measure.
Time Frame: Baseline, Weeks 1, 2, 3, 8, 16, 24, and 48
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 44 | 43
pg/mL
  Baseline (n=44, 42) | 37.61 (11.12) | 39.39 (10.16)
  Week 1: Absolute values (n=44, 43) | 51.03 (59.12) | 237.34 (71.38)
  Week 1: Change From Baseline (n=44, 42) | 13.42 (57.91) | 198.39 (69.41)
  Week 2: Absolute values (n=43, 41) | 44.07 (42.15) | 329.90 (81.93)
  Week 2: Change From Baseline (n=43, 40) | 6.13 (41.60) | 291.38 (79.29)
  Week 3: Absolute values (n=44, 40) | 41.64 (27.07) | 384.88 (99.41)
  Week 3: Change From Baseline (n=44, 39) | 4.03 (26.00) | 346.68 (95.96)
  Week 8: Absolute values (n=42, 39) | 38.66 (11.95) | 486.62 (116.41)
  Week 8: Change From Baseline (n=42, 38) | 0.91 (5.07) | 447.77 (114.40)
  Week 16: Absolute values (n=32, 33) | 37.71 (10.30) | 525.48 (164.90)
  Week 16: Change From Baseline (n=32, 32) | -0.08 (5.71) | 486.43 (163.32)
  Week 24: Absolute values (n=36, 34) | 38.72 (13.06) | 520.18 (167.97)
  Week 24: Change From Baseline (n=36, 33) | 1.11 (6.47) | 482.10 (168.44)
  Week 48: Absolute values (n=32, 27) | 36.52 (9.93) | 491.44 (164.82)
  Week 48: Change From Baseline (n=32, 26) | -0.75 (5.20) | 454.19 (163.93)

15. Secondary Outcome: Percentage of Participants With Anti-Tocilizumab Antibody
Time Frame: Baseline, and post-baseline (up to Week 48)
Population: Safety population. Here, number of participants analyzed included only those participants who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Tocilizumab
Number analyzed (Participants) | 43 | 42
percentage of participants
  Baseline | 7.0 | 2.4
  Post-Baseline | 0.0 | 2.4

ADVERSE EVENTS:
Time Frame: Up to Week 96 (reporting groups up to 24 Weeks and up to 48 Weeks present data as of the 11 July 2014 data cut-off date; reporting groups up to 96 weeks present data as of the 05 August 2015 data cut-off date).
Description: MedDRA 17.0 was utilized up to Week 48; MedDRA 18.0 was utilized for Week 48 up to Week 96
Groups:
- Placebo (up to 24 Weeks): Participants received TCZ matched placebo by SC injection qw for Week 0 to Week 48 (blinded-treatment period) and then received TCZ (162 mg) SC injection qw in the open-label period for Week 48 to Week 96. The data analyzed for placebo up to Week 24 are presented in this reporting group.
- Tocilizumab (up to 24 Weeks): Participants received TCZ (162 mg) by SC injection qw for Week 0 to Week 48 (blinded-treatment period) and then in the open-label period for Week 48 to Week 96. The data analyzed for TCZ up to Week 24 was presented in this reporting group.
- Placebo (up to 48 Weeks): Participants received TCZ matched placebo by SC injection qw for Week 0 to Week 48 (blinded-treatment period) and then received TCZ (162 mg) SC injection qw in the open-label period for Week 48 to Week 96. The data analyzed for placebo up to Week 48 are presented in this reporting group.
- Tocilizumab (up to 48 Weeks): Participants received TCZ (162 mg) by SC injection qw for Week 0 to Week 48 (blinded-treatment period) and then in the open-label period for Week 48 to Week 96. The data analyzed for TCZ up to Week 48 are presented in this reporting group.
- Placebo to Tocilizumab (up to 96 Weeks): Participants received TCZ matched placebo by SC injection qw for Week 0 to Week 48 (blinded-treatment period) and then received TCZ (162 mg) SC injection qw in the open-label period for Week 48 to Week 96. The data analyzed for double-blind placebo to open-label tocilizumab up to Week 96 are presented in this reporting group.
- Tocilizumab to Tocilizumab (up to 96 Weeks): Participants received TCZ (162 mg) by SC injection qw for Week 0 to Week 48 (blinded-treatment period) and then in the open-label period for Week 48 to Week 96. The data analyzed for double-blind tocilizumab to open-label tocilizumab up to Week 96 are presented in this reporting group.
Arm/Group | Placebo (up to 24 Weeks) | Tocilizumab (up to 24 Weeks) | Placebo (up to 48 Weeks) | Tocilizumab (up to 48 Weeks) | Placebo to Tocilizumab (up to 96 Weeks) | Tocilizumab to Tocilizumab (up to 96 Weeks)
Serious Adverse Events (participants affected / at risk) | 11/44 | 9/43 | 15/44 | 14/43 | 22/44 | 17/43
Other Adverse Events (participants affected / at risk) | 26/44 | 28/43 | 32/44 | 34/43 | 39/44 | 38/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (up to 24 Weeks) (N=44) | Tocilizumab (up to 24 Weeks) (N=43) | Placebo (up to 48 Weeks) (N=44) | Tocilizumab (up to 48 Weeks) (N=43) | Placebo to Tocilizumab (up to 96 Weeks) (N=44) | Tocilizumab to Tocilizumab (up to 96 Weeks) (N=43)
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0
Cyanosis (Cardiac disorders) | 1 | 0 | 1 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Retroperitoneal fibrosis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0
Impaired healing (General disorders) | 0 | 1 | 0 | 1 | 0 | 1
Multi-organ failure (General disorders) | 0 | 0 | 0 | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1 | 0 | 1 | 2 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 2 | 1 | 2 | 2 | 2
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Post procedural cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Systemic sclerosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 — The previous event Renal failure acute at Week 48 was updated to Acute kidney injury at Week 96
Scleroderma renal crisis (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 2 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 2 | 1 | 2
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 1
Hypertensive emergency (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Autoimmune thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (up to 24 Weeks) (N=44) | Tocilizumab (up to 24 Weeks) (N=43) | Placebo (up to 48 Weeks) (N=44) | Tocilizumab (up to 48 Weeks) (N=43) | Placebo to Tocilizumab (up to 96 Weeks) (N=44) | Tocilizumab to Tocilizumab (up to 96 Weeks) (N=43)
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 0 | 0 | 2 | 4 — One case of abdominal pain was updated between Week 24 and 48 to diverticulum. The remaining 2 cases at week 48 fall below the 5% threshold and are therefore not presented.
Diarrhoea (Gastrointestinal disorders) | 4 | 6 | 4 | 7 | 5 | 12
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 3 | 3 | 3 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 4 | 5 | 5 | 7 | 5
Nausea (Gastrointestinal disorders) | 0 | 0 | 3 | 2 | 5 | 3
Vomiting (Gastrointestinal disorders) | 0 | 3 | 1 | 3 | 2 | 3
Asthenia (General disorders) | 3 | 0 | 3 | 0 | 3 | 0
Fatigue (General disorders) | 2 | 4 | 2 | 5 | 3 | 6
Oedema peripheral (General disorders) | 1 | 3 | 1 | 3 | 3 | 4
Herpes zoster (Infections and infestations) | 0 | 0 | 2 | 3 | 2 | 4
Infected skin ulcer (Infections and infestations) | 5 | 0 | 5 | 1 | 7 | 3
Nasopharyngitis (Infections and infestations) | 2 | 3 | 4 | 5 | 5 | 8
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 6 | 1 | 8 | 3
Urinary tract infection (Infections and infestations) | 3 | 2 | 3 | 3 | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 6 | 8 | 6 | 10 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5 | 3 | 6 | 3 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 5 | 2 | 5 | 2 | 7
Dizziness (Nervous system disorders) | 2 | 3 | 2 | 3 | 2 | 5
Headache (Nervous system disorders) | 2 | 3 | 3 | 5 | 5 | 8
Sleep disorder (Psychiatric disorders) | 0 | 0 | 3 | 1 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 3 | 4 | 3 | 5 — The Investigator removed an adverse event of dyspnoea between Week 24 and Week 48 reporting events.
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 7 | 4 | 8 | 9 | 12
Skin ulcer (Skin and subcutaneous tissue disorders) | 6 | 6 | 7 | 7 | 9 | 8
Hypertension (Vascular disorders) | 0 | 0 | 3 | 2 | 4 | 3
Raynaud's phenomenon (Vascular disorders) | 1 | 3 | 2 | 5 | 2 | 6
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 2
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 2
Injection site erythema (General disorders) | 0 | 0 | 0 | 0 | 2 | 3
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 3 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 3
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.